CLINICAL TRIAL: NCT05030558
Title: Effect of Web Supported Interactive Nursing Program on Illness Perception, Pain Management and Disease Intensity in Fibromyalgia: A Mixed Method Study
Brief Title: Web-supported Interactive Nurse Program in Fibromyalgia Patients: A Mixed Method Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meryem Otu (Other)
Collaborators: Cumhuriyet University (Other)
Responsible Party: Sponsor-Investigator, Meryem Otu, Nurse, Cumhuriyet University
Organization: Cumhuriyet University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Sivas Cumhuriyet University
Record Dates: First submitted 2021-08-25; First posted 2021-09-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Web based intervention; Nursing; Illness perception
MeSH Terms: conditions — Fibromyalgia | interventions — Growth Differentiation Factor 15

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant
Masking Description: Patients participating in the study will know that they are in a randomized controlled study, but they will not know which group they are in until the study is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): The web-supported interactive nursing program intervention will last 4 weeks. In the first week of the training, the identity and causes of the disease, which is one of the sub-dimensions of the perception of illness, will be emphasized, and the themes of misperception determined in this field through qualitative study will be emphasized. In the second week, they will be asked to look at training sessions that discuss perceptions of the illness's timeline and consequences. In the last two weeks of the training, they will be asked to attend the trainings for the control of Fibromyalgia symptoms. During the study, short mobile phone messages containing reminders and motivations will be sent regularly twice a week (8 times). Data collection forms will be applied to the intervention group 3 times before starting the web-based interactive nurse program, at the end of the program (in the 1st month) and then at the end of the 2nd month.
  Interventions: Behavioral: Web-assisted patient education intervention designed according to the common-sense model
- Control Group (Active Comparator): The Fibromyalgia patient booklet of the Turkish Physical Medicine and Rehabilitation Association will be available in pdf format on the website of the participants assigned to the control group. Participants in this group will be able to access other trainings after the end of the study, if they wish.
  Data collection forms will be applied to the control group 3 times in total, before the start of the study, in the 1st month and the 2nd month of the study.
  Interventions: Behavioral: The website where the Turkish Physical Medicine and Rehabilitation Association Fibromyalgia patient booklet is available as pdf.

INTERVENTIONS:
Behavioral: Web-assisted patient education intervention designed according to the common-sense model — Implementation of patient education with the website created about fibromyalgia disease in 4 weeks according to the disease perception themes reached as a result of the qualitative research.
  Arms: Interventional group
Behavioral: The website where the Turkish Physical Medicine and Rehabilitation Association Fibromyalgia patient booklet is available as pdf. — The website where the Turkish Physical Medicine and Rehabilitation Association Fibromyalgia patient booklet is available as pdf.
  Arms: Control Group

SUMMARY:
This study was planned to examine the effect of the web-supported interactive nurse program developed in line with the Common-Sense Model on the perception of illness, coping with pain and severity of illness in fibromyalgia patients. Mixed method is a research. The exploratory sequential design, one of the mixed research methods, will be used. The research will continue with the quantitative part starting with the qualitative part. The quantitative part of the research is a randomized controlled experimental study.

DETAILED DESCRIPTION:
Fibromyalgia is a very common musculoskeletal disease characterized by increased pain sensitivity. Hospital admissions are increasing with symptoms such as fibromyalgia, chronic pain, fatigue, sleep disturbance, depression and cognitive problems, and this is reflected in general health care expenditures. The absence of objective markers to diagnose the disease, the social recognition of fibromyalgia, and the negative perception of the disease by patients in its clinical management creates a permanent problem. Individuals who perceive fibromyalgia as having more severe cognitive consequences and less controllable are more affected by the symptoms of the disease. Therefore, understanding the patient's perceptions of the disease is important for effective health management and reducing the severity of the disease and improving the patient's health outcomes. Although there are many descriptive studies showing that fibromyalgia patients have a negative perception of illness, no study has been found in which the effectiveness of the education offered with the self-regulation model for the perception of illness was evaluated in fibromyalgia patients.

Aim: This research was planned to examine the effect of the Web-Assisted Interactive Nursing Program designed according to the Common-Sense Model on the perception of illness, coping with pain and severity of illness in fibromyalgia patients.

Method: The study was designed as an exploratory mixed method research in which qualitative and quantitative research methods were used together. The qualitative and quantitative research sample will consist of patients diagnosed with fibromyalgia according to the American College of Rheumatology (ACR) 2010 Criteria by the physician. "Criteria sampling method", one of the purposive sampling methods used in qualitative research, will be used to determine the individuals to be included in the qualitative part of the research. Qualitative interviews will be conducted face to face. Interviews with people will continue until data saturation is reached. In the qualitative part of the research, individual in-depth interview method will be selected and "Semi-Structured Interview Form" will be used as a data collection tool. Interviews with people will continue until data saturation is reached. All interviews will be recorded in digital format, transcribed and then transferred to the qualitative analysis software MAXQDA. In line with the data obtained in the qualitative dimension of the research, the design of the web-supported interactive nursing program will be created.

The quantitative part of the study will be carried out as a randomized controlled trial using the block randomization method. Randomization will be done by a statistician other than the researcher. Power analysis was calculated using G * Power 3.1.9.7 program. With 0.95 effect size, 95% power and 0.05 significance level, the required sample size was determined as 30 individuals per group, and 60 individuals in total. It was decided to include 70 individuals, 35 individuals in the intervention group and 31 individuals in the control group, by taking 15% more of the calculated sample against the possibility of sample loss during the study. In the quantitative part of the research, the web-supported interactive nurse program will last 1 month and the application will last for 2 months. A text message will be sent to their phone to remind individuals to use the website. Messages will be sent twice a week, for a total of 8 times. Visual Analogue Scale (VAS), Website Usability Scale, Illness Perception Scale (IPQ), Pain Coping Scale (PCI), Fibromyalgia Impact Questionnaire (FIQ) will be used as measurement tools. Data collection forms will be applied to the intervention and control groups three times in total, before the start of the WeB-supported interactive nurse program, at the end of the Web-supported interactive nurse program (1st month) and at the 2nd month. The data obtained after each evaluation will be transferred to the "Statistical Package for Social Sciences Software" (SPSS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a mean score of 4 or greater on the Visual Analogue Scale (VAS)
* Patients whose drug treatment was stable and no non-pharmacological intervention was applied during the study period,
* Patients with basic computer literacy,
* Patients with computer access.

Exclusion Criteria:

* Individuals with secondary inflammatory rheumatic disease or another diagnosed disease that may contribute to chronic pain
* Patients with hearing, vision and understanding problems,
* Patients whose drug therapy was changed or who received any non-pharmacological therapy during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Before application
  VAS provides rapid measurement of pain intensity in clinical and laboratory conditions. In VAS, the patient is asked to make a mark on a 10 cm horizontal line showing the current situation. In this study, for pain; Markings are made on a 10 cm horizontal line, one end of which indicates the patient's pain is very good (0 = no pain) and the other end is very bad (10 = most severe).
Visual Analog Scale | Immediately after application (1st mounth)
  VAS provides rapid measurement of pain intensity in clinical and laboratory conditions. In VAS, the patient is asked to make a mark on a 10 cm horizontal line showing the current situation. In this study, for pain; Markings are made on a 10 cm horizontal line, one end of which indicates the patient's pain is very good (0 = no pain) and the other end is very bad (10 = most severe).
Visual Analog Scale | 1 month after application (2nd mounth)
  VAS provides rapid measurement of pain intensity in clinical and laboratory conditions. In VAS, the patient is asked to make a mark on a 10 cm horizontal line showing the current situation. In this study, for pain; Markings are made on a 10 cm horizontal line, one end of which indicates the patient's pain is very good (0 = no pain) and the other end is very bad (10 = most severe).
Illness Perception Scale | Before application
  The scale consists of 70 items and three sub-dimensions:
  * Type of disease,
  * Opinions about the disease,
  * Dimensions of disease causes. Disease Type Dimension: It consists of 14 items. It is answered with yes or no. The sum of yes answers gives the score for this sub-dimension. Opinions on the Disease Dimension: This sub-dimension consists of 38 items. Responses to each item are evaluated with a five-point Likert-type measurement ranging from "1: I definitely don't think" to "5: I definitely think". Causes of Disease Dimension: It consists of 18 items that investigate the patient's thoughts about the possible causes of the disease. A five-point Likert type measurement is used. The score of the entire scale is found by summing the scores obtained from these sub-dimensions.
Illness Perception Scale | Immediately after application (1st mounth)
  The scale consists of 70 items and three sub-dimensions:
  * Type of disease,
  * Opinions about the disease,
  * Dimensions of disease causes. Disease Type Dimension: It consists of 14 items. It is answered with yes or no. The sum of yes answers gives the score for this sub-dimension. Opinions on the Disease Dimension: This sub-dimension consists of 38 items. Responses to each item are evaluated with a five-point Likert-type measurement ranging from "1: I definitely don't think" to "5: I definitely think". Causes of Disease Dimension: It consists of 18 items that investigate the patient's thoughts about the possible causes of the disease. A five-point Likert type measurement is used. The score of the entire scale is found by summing the scores obtained from these sub-dimensions.
Illness Perception Scale | 1 month after application (2nd mounth)
  The scale consists of 70 items and three sub-dimensions:
  * Type of disease,
  * Opinions about the disease,
  * Dimensions of disease causes. Disease Type Dimension: It consists of 14 items. It is answered with yes or no. The sum of yes answers gives the score for this sub-dimension. Opinions on the Disease Dimension: This sub-dimension consists of 38 items. Responses to each item are evaluated with a five-point Likert-type measurement ranging from "1: I definitely don't think" to "5: I definitely think". Causes of Disease Dimension: It consists of 18 items that investigate the patient's thoughts about the possible causes of the disease. A five-point Likert type measurement is used. The score of the entire scale is found by summing the scores obtained from these sub-dimensions.
Pain Coping Questionnaire | Before application
  The scale evaluates chronic pain patients' ways of coping with organic or psychogenic pain. The 29-item self-report scale is answered on a 4-point Likert scale (0 = never, 3 = often). Scores range from 0 to 3 for each item. The total score for each subtest is calculated by summing the scores obtained from the items in that subtest.
Pain Coping Questionnaire | Immediately after application (1st mounth)
  The scale evaluates chronic pain patients' ways of coping with organic or psychogenic pain. The 29-item self-report scale is answered on a 4-point Likert scale (0 = never, 3 = often). Scores range from 0 to 3 for each item. The total score for each subtest is calculated by summing the scores obtained from the items in that subtest.
Pain Coping Questionnaire | 1 month after application (2nd mounth)
  The scale evaluates chronic pain patients' ways of coping with organic or psychogenic pain. The 29-item self-report scale is answered on a 4-point Likert scale (0 = never, 3 = often). Scores range from 0 to 3 for each item. The total score for each subtest is calculated by summing the scores obtained from the items in that subtest.
Fibromyalgia Impact Questionnaire | Before application
  The scale measures 10 different characteristics: physical function, well-being, absenteeism, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. Higher scores indicate that the disease affects the person more. The total score can be between 0-80. A score of 80 indicates high influence.
Fibromyalgia Impact Questionnaire | Immediately after application (1st mounth)
  The scale measures 10 different characteristics: physical function, well-being, absenteeism, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. Higher scores indicate that the disease affects the person more. The total score can be between 0-80. A score of 80 indicates high influence.
Fibromyalgia Impact Questionnaire | 1 month after application (2nd mounth)
  The scale measures 10 different characteristics: physical function, well-being, absenteeism, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. Higher scores indicate that the disease affects the person more. The total score can be between 0-80. A score of 80 indicates high influence.

SECONDARY OUTCOMES:
Website Usability Scale | Immediately after application (1st mounth)
  The scale consists of a total of 25 questions with four sub-dimensions (ease of navigation = 10 questions, design = 7 questions, ease of access = 4 questions, ease of use = 4 questions). The answers to the items of the scale are collected with a Likert-type five-point rating scale. The scale consists of "Strongly agree (5)", "Agree (4)", "Undecided (3)", "Disagree (2)" and "Strongly disagree (1)". 21 of the items in the scale are positive and 4 of them are negative items. The lowest score to be taken from the scale is 25 and the highest score is 125.

CONTACTS AND LOCATIONS:
Overall Officials: Şerife Karagözoğlu, Prof. Dr., Study Director — Cumhuriyet University
Locations (1):
- Meryem Otu, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No